CLINICAL TRIAL: NCT02788279
Title: A Phase III, Open-Label, Multicenter, Three-Arm, Randomized Study to Investigate the Efficacy and Safety of Cobimetinib Plus Atezolizumab and Atezolizumab Monotherapy vs. Regorafenib in Patients With Previously Treated Unresectable Locally Advanced or Metastatic Colorectal Adenocarcinoma
Brief Title: A Study to Investigate Efficacy and Safety of Cobimetinib Plus Atezolizumab and Atezolizumab Monotherapy Versus Regorafenib in Participants With Metastatic Colorectal Adenocarcinoma (COTEZO IMblaze370)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO30182; 2016-000202-11 (EudraCT Number)
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Cancer
Keywords: Locally advanced or Metastatic colorectal adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; cobimetinib; regorafenib

ARMS (3):
- Atezolizumab (Experimental): Participants will receive atezolizumab monotherapy 1200 milligrams (mg) intravenous (IV) on Day 1 in a 21-day cycle until disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PDL1 Antibody
- Cobimetinib + Atezolizumab (Experimental): Participants will receive cobimetinib 60 mg orally on Days 1 to 21 plus atezolizumab 840 mg IV on Day 1 and Day 15 in a 28-day cycle until disease progression according to RECIST Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PDL1 Antibody; Drug: Cobimetinib
- Regorafenib (Active Comparator): Participants will receive regorafenib 160 mg orally on Days 1 to 21 in a 28-day cycle until disease progression according to RECIST Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an Engineered Anti-PDL1 Antibody — Participants will receive atezolizumab IV at 840 mg on Day 1 and Day 15 in a 28-day cycle as a combination therapy or at 1200 mg on Day 1 in a 21-day cycle as a monotherapy until disease progression according to RECIST Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
  Arms: Atezolizumab; Cobimetinib + Atezolizumab
Drug: Cobimetinib — Participants will receive cobimetinib 60 mg orally on Days 1 to 21 in a 28-day cycle as a combination therapy until disease progression according to RECIST Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
  Arms: Cobimetinib + Atezolizumab
Drug: Regorafenib — Participants will receive regorafenib 160 mg orally on Days 1 to 21 in a 28-day cycle until disease progression according to RECIST Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
  Arms: Regorafenib

SUMMARY:
This is a Phase III, multicenter, open-label, three-arm, randomized study in participants with unresectable locally advanced or metastatic colorectal cancer (CRC) who have received at least two prior regimens of cytotoxic chemotherapy for metastatic disease. The study compares regorafenib, a standard of care therapy in this setting, to cobimetinib plus atezolizumab and atezolizumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

Disease-specific inclusion criteria:

* Histologically confirmed adenocarcinoma originating from the colon or rectum (Stage 4 American Joint Committee on Cancer [AJCC] 7th edition)
* Experienced disease progression or was intolerant to at least two systemic chemotherapy regimens for metastatic colorectal cancer that must have included fluroropyrimidines, irinotecan, and oxaliplatin; adjuvant regimen can be considered as one chemotherapy regimen for metastatic disease if the participant had disease recurrence within 6 months of completion; disease progression must have occurred within 3 months of the last systemic therapy administration

General inclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Anticipated life expectancy greater than or equal to (>=) 3 months
* Adequate hematologic and end organ function
* Women of childbearing potential must agree to appropriately use an effective form of contraception (failure rate of less than [<] 1 percent [%] per year) during the treatment period, within 5 months after the last dose of atezolizumab, and within 3 months after the last dose of cobimetinib and regorafenib
* Men must agree not to donate sperm or have intercourse with a female partner without using appropriate barrier contraception during the treatment period and for 3 months after the last dose of either cobimetinib or regorafenib
* Provide an archival or newly obtained tumor tissue sample

Exclusion Criteria:

* After the approximate 5% cap for microsatellite (MSI)-high participants is reached, only MSI-stable participants will be eligible
* Once the 50% cap for wild-type RAS has been reached, only extended RAS-mutant participants will be eligible
* Major surgery or radiotherapy within 21 days prior to Cycle 1 Day 1 or anticipation of needing such procedure while receiving study treatment
* Treatment with any anti-cancer agent within 14 days prior to Cycle 1 Day 1
* Uncontrolled tumor-related pain. Participants requiring narcotic pain medication must be on a stable regimen at study entry
* Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage more than once every 28 days. Indwelling drainage catheters (e.g., PleurX®) are allowed
* Active or untreated central nervous system (CNS) metastases are excluded
* Prior therapy with any cancer immunotherapy, MEK inhibitor, or regorafenib
* Participants with active malignancy (other than CRC) or a prior malignancy within the past 3 years are excluded. Participants with completely resected cutaneous melanoma (early stage), basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in-situ, breast carcinoma in-situ, and localized prostate cancer are eligible
* Unstable angina, new onset angina within last 3 months, myocardial infarction within last 6 months and current congestive heart failure New York Heart Association Class II or higher
* Left ventricular ejection fraction (LVEF) below institutional lower limit of normal or below 50%, whichever is lower
* Poorly controlled hypertension, defined as a blood pressure consistently above 150/90 millimeters of Mercury (mmHg) despite optimal medical management
* Human immunodeficiency virus (HIV) infection
* Active tuberculosis infection
* Severe infections within 2 weeks prior to Cycle 1 Day 1
* Active or chronic viral hepatitis B or C infection
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for central serous retinopathy, retinal vein occlusion, or neovascular macular degeneration
* Participants will be excluded if they currently have any of the risk factors as defined in the study protocol for retinal vein occlusion
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, bronchiolitis obliterans, drug-induced pneumonitis, or idiopathic pneumonitis
* History of organ transplantation including allogeneic bone marrow transplantation
* Inability to swallow medications
* Malabsorption condition that would alter the absorption of orally administered medications
* Pregnant, lactating, breastfeeding, or intending to become pregnant during the study
* Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation of a live attenuated vaccine will be required during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (73):
- United States (17):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Florida Cancer Specialists; SCRI, Fort Myers, Florida
  - Cancer Specialists; North Florida ;Jacksonville (AC Skinner Pkwy), Jacksonville, Florida
  - Florida Cancer Specialists., St. Petersburg, Florida
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Southdale Cancer Clinic U of M Medical Center, Fairview- Edina, Edina, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - North Shore Hem Onc Associates, East Setauket, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - INTEGRIS Cancer Inst of OK, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute; Division of Medical Oncology, Pittsburgh, Pennsylvania
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Medical Oncology Associates, Spokane, Washington
- Australia (6):
  - Port Macquarie Base Hospital;North Coast Cancer Institute, Port Macquarie, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Sydney Adventist Hospital; Clinical Trial Unit, Sydney, New South Wales
  - Monash Medical Centre; Oncology, Clayton, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Austin Health; Cancer Clinical Trial Centre, Heidelberg, Victoria
- Belgium (5):
  - Imeldaziekenhuis, Bonheiden
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Notre Dame, Charleroi
  - AZ Groeninge, Kortrijk
  - UZ Leuven Gasthuisberg, Leuven
- Canada (8):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - Cross Cancer Institute; Clinical Trials, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - McGill University Health Center, Cedar Cancer Center, Montreal, Quebec
  - Hopital du Sacre-Coeur, Montreal, Quebec
  - CHU de Québec, Québec, Quebec
- Hong Kong (3):
  - Queen Mary Hospital; Dept. of Clinical Oncology, Hong Kong
  - Tuen Mun Hospital; Clinical Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- Italy (7):
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Oncologia, San Giovanni Rotondo, Apulia
  - Azienda Osp Uni Seconda Università Degli Studi Di Napoli; Unità Operativa Oncologia Medica, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena; Oncologia, Modena, Emilia-Romagna
  - Istit. Naz. per la Ricerca sul Cancro - Az. Osped. S. Martino, Genoa, Liguria
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - A.O. Universitaria Pisana; Oncologia, Pisa, Tuscany
- Poland (5):
  - Centrum Onkologii im. Prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne; Klinika Onkologii i Radioterapii, Gdansk
  - Szpitale Pomorskie Sp. z o. o., Gdynia
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - Woj.Wielospecjalistyczne Centrum Onkologii i Traumatologii; Oddz.Hematologii Pododz.Chemioterapii, Lodz
- Russia (3):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - N.N.Burdenko Main Military Clinical Hospital; Oncology Dept, Moscow
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
- South Korea (6):
  - National Cancer Center, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Health System/Severance Hospital, Seoul
- Spain (6):
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Clínico Universitario de Valencia; Servicio de Oncología, Valencia
- United Kingdom (7):
  - Birmingham Heartlands Hospital; Dept of Oncology, Birmingham
  - Royal Marsden Hospital - Fulham; Oncology Department, London
  - The Christie; GI Research Office, Manchester
  - Churchill Hospital; Department of Oncology, Oxford
  - Queen's Hospital, Romford
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton

REFERENCES:
- [Derived] Taraborrelli L, Senbabaoglu Y, Wang L, Lim J, Blake K, Kljavin N, Gierke S, Scherl A, Ziai J, McNamara E, Owyong M, Rao S, Calviello AK, Oreper D, Jhunjhunwala S, Argiles G, Bendell J, Kim TW, Ciardiello F, Wongchenko MJ, de Sauvage FJ, de Sousa E Melo F, Yan Y, West NR, Murthy A. Tumor-intrinsic expression of the autophagy gene Atg16l1 suppresses anti-tumor immunity in colorectal cancer. Nat Commun. 2023 Sep 23;14(1):5945. doi: 10.1038/s41467-023-41618-7. PMID 37741832
- [Derived] Barteselli G, Goodman GR, Patel Y, Caro I, Xue C, McCallum S. Characterization of Serous Retinopathy Associated with Cobimetinib: Integrated Safety Analysis of Four Studies. Drug Saf. 2022 Dec;45(12):1491-1499. doi: 10.1007/s40264-022-01248-2. Epub 2022 Oct 30. PMID 36310331
- [Derived] Eng C, Kim TW, Bendell J, Argiles G, Tebbutt NC, Di Bartolomeo M, Falcone A, Fakih M, Kozloff M, Segal NH, Sobrero A, Yan Y, Chang I, Uyei A, Roberts L, Ciardiello F; IMblaze370 Investigators. Atezolizumab with or without cobimetinib versus regorafenib in previously treated metastatic colorectal cancer (IMblaze370): a multicentre, open-label, phase 3, randomised, controlled trial. Lancet Oncol. 2019 Jun;20(6):849-861. doi: 10.1016/S1470-2045(19)30027-0. Epub 2019 Apr 16. PMID 31003911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 490 participants were screened of whom only 363 participants were randomized.
Groups:
- Regorafenib: Participants received regorafenib 160 milligrams (mg) orally once daily on Days 1 to 21 in a 28-day cycle until disease progression according to RECIST Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
- Cobimetinib + Atezolizumab: Participants received cobimetinib 60 mg orally on Days 1 to 21 plus atezolizumab 840 mg IV on Day 1 and Day 15 in a 28-day cycle until disease progression according to RECIST Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
- Atezolizumab: Participants received atezolizumab monotherapy 1200 mg intravenous (IV) on Day 1 in a 21-day cycle until disease progression according to RECIST Version 1.1, unacceptable toxicity, death, participant's or physician decision to withdraw, or pregnancy, whichever occurs first.
Period: Overall Study
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
Started (Intent to treat (ITT) population) | 90 | 183 | 90
Received Treatment (Safety Population) | 80 | 179 | 90
Modified ITT Population (Patient-reported outcome (PRO)) | 57 | 125 | 61
Completed | 0 | 0 | 0
Not Completed | 90 | 183 | 90
Not completed — Death | 62 | 136 | 72
Not completed — Withdrawal by Subject | 10 | 15 | 5
Not completed — Lost to Follow-up | 0 | 3 | 2
Not completed — Sponsor decision | 18 | 29 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab | Total
Number analyzed (Participants) | 90 | 183 | 90 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (10.3) | 58.0 (11.9) | 56.7 (10.2) | 57.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 75 | 31 | 145
  Male | 51 | 108 | 59 | 218
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 5 | 25
  Not Hispanic or Latino | 77 | 166 | 82 | 325
  Unknown or Not Reported | 4 | 6 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 12 | 18 | 11 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 0 | 8 | 2 | 10
  White | 71 | 152 | 73 | 296
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 4 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time (in months) between the date of randomization and the date of death due to any cause. Participants who were not reported as having died at the date of analysis were censored at the date when they were last known to be alive. Participants who did not have post-baseline information were censored at the date of randomization + 1 day. Median OS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley.
Time Frame: From randomization up to death due to any cause (up to approximately 20 months)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
Number analyzed (Participants) | 90 | 183 | 90
months | 8.51 [6.41 to 10.71] | 8.87 [7.00 to 10.61] | 7.10 [6.05 to 10.05]
Statistical Analysis 1: Comparison: Regorafenib vs Cobimetinib + Atezolizumab; Test type: Superiority; p = 0.9871, Stratified Log-Rank; Stratification factors included extended RAS mutation status and time since diagnosis of first metastasis; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.73 to 1.38] — Hazard ratio was estimated using stratified Cox regression
Statistical Analysis 2: Comparison: Regorafenib vs Atezolizumab; Test type: Superiority; p = 0.3360, Stratified Log-Rank; Stratification factors included extended RAS mutation status and time since diagnosis of first metastasis; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.83 to 1.71] — Hazard ratio was estimated using stratified Cox regression
Statistical Analysis 3: Comparison: Regorafenib vs Cobimetinib + Atezolizumab; Test type: Superiority; p = 0.9686, Unstratified Log-Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.74 to 1.38] — Hazard ratio was estimated using unstratified Cox regression
Statistical Analysis 4: Comparison: Regorafenib vs Atezolizumab; Test type: Superiority; p = 0.3553, Unstratified Log-Rank; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.83 to 1.69] — Hazard ratio was estimated using unstratified Cox regression

2. Secondary Outcome: Progression-Free Survival (PFS) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: PFS was defined as the time from randomization to disease progression as determined by the investigator with the use of RECIST v1.1 or death due to any cause, whichever occurred earlier. Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). For non-target lesions, disease progression was defined as unequivocal progression of existing lesions. The appearance of one or more new lesions was also considered progression. Participants who did not have post-baseline information were censored at the date of randomization + 1 day. Median OS was estimated by Kaplan-Meier method and 95% CI was assessed using the method of Brookmeyer and Crowley.
Time Frame: From randomization up to disease progression or death due to any cause (up to approximately 20 months)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
Number analyzed (Participants) | 90 | 183 | 90
months | 2.00 [1.87 to 3.61] | 1.91 [1.87 to 1.97] | 1.94 [1.91 to 2.10]
Statistical Analysis 1: Comparison: Regorafenib vs Cobimetinib + Atezolizumab; Test type: Superiority; p = 0.1208, Stratified Log-Rank; Stratification factors included extended RAS mutation status and time since diagnosis of first metastasis; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.94 to 1.65] — Hazard ratio was estimated using stratified Cox regression
Statistical Analysis 2: Comparison: Regorafenib vs Atezolizumab; Test type: Superiority; p = 0.0509, Stratified Log-Rank; Stratification factors included extended RAS mutation status and time since diagnosis of first metastasis; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [1.00 to 1.94] — Hazard ratio was estimated using stratified Cox regression
Statistical Analysis 3: Comparison: Regorafenib vs Cobimetinib + Atezolizumab; Test type: Superiority; p = 0.1726, Unstratified Log-Rank; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.92 to 1.60] — Hazard ratio was estimated using unstratified Cox regression
Statistical Analysis 4: Comparison: Regorafenib vs Atezolizumab; Test type: Superiority; p = 0.0467, Unstratified Log-Rank; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [1.00 to 1.91] — Hazard ratio was estimated using unstratified Cox regression

3. Secondary Outcome: Percentage of Participants With Investigator-Assessed Objective Response of Complete Response (CR) or Partial Response (PR) According to RECIST Version 1.1
Description: PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker levels (as applicable to non-target lesions). Objective response and its 95% CI were calculated using the Clopper-Pearson method.
Time Frame: From randomization up to death due to any cause (up to approximately 20 months)
Population: Analysis was performed on evaluable participants in the ITT population with measurable disease at baseline, as determined by the investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
Number analyzed (Participants) | 90 | 183 | 90
percentage of participants | 2.2 [0.27 to 7.80] | 2.7 [0.89 to 6.26] | 2.2 [0.27 to 7.80]
Statistical Analysis 1: Comparison: Regorafenib vs Cobimetinib + Atezolizumab; Test type: Superiority; p = 1.0000, Stratified Cochrane-Mantel-Haenszel; Stratification factors included extended RAS mutation status and time since diagnosis of first metastasis; Difference in Response Rates = 0.51, 95% CI 2-sided [-3.92 to 4.94] — 95% CI for difference in response rates was constructed using Hauck-Anderson method
Statistical Analysis 2: Comparison: Regorafenib vs Atezolizumab; Test type: Superiority; p = 1.0000, Stratified Cochran-Mantel-Haenszel; Stratification factors included extended RAS mutation status and time since diagnosis of first metastasis; Difference in Response Rates = 0.00, 95% CI 2-sided [-4.89 to 4.89] — 95% CI for difference in response rates was constructed using Hauck-Anderson method

4. Secondary Outcome: Duration of Response (DOR) According to RECIST Version 1.1
Description: DOR is defined as the period measured from the date of the first occurrence of a CR or PR (whichever status is recorded first) until the first date that progressive disease or death is documented. Disease progression was determined on the basis of investigator assessment with use of RECIST v1.1. Median DOR was estimated using the Kaplan-Meier method, and the 95% CI was calculated using the method of Brookmeyer and Crowley.
Time Frame: From first occurrence of CR or PR up to disease progression or death due to any cause (up to approximately 20 months)
Population: DOR was assessed in participants who had an objective response during the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
Number analyzed (Participants) | 2 | 5 | 2
months | 4.50 [3.61 to 5.39] | 1.97 [1.77 to 3.81] | 2.81 [1.84 to 3.78]

5. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life-C30 Questionnaire (EORTC QLQ-C30) Physical Functioning Sub-scale Score
Description: The EORTC QLQ-C30 questionnaire consisted of 30 questions generating five functional scores (physical, role, cognitive, emotional, and social); a global health status/global quality of life scale score; three symptom scale scores (fatigue, pain, and nausea and vomiting); and six stand alone one-item scores that capture additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and perceived financial burden. All the scales and single-item scores were linearly transformed so that each score ranged from 0 to 100. A higher score on the global health and functioning subscales is indicative of better functioning.
Time Frame: Baseline, end of the study (up to approximately 2.5 years)
Population: Analysis was performed on PRO-evaluable population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'Number Analyzed' signifies the number of participants evaluable at specified time point.
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
Number analyzed (Participants) | 57 | 125 | 61
units of a scale
  Week 3: number analyzed (Participants) | 0 | 0 | 49
  Week 3 |  |  | -1.50 (10.56)
  Week 4: number analyzed (Participants) | 44 | 100 | 0
  Week 4 | -6.52 (13.90) | -3.92 (11.05) |
  Week 6: number analyzed (Participants) | 0 | 0 | 48
  Week 6 |  |  | -0.14 (12.49)
  Week 8: number analyzed (Participants) | 29 | 78 | 0
  Week 8 | -8.97 (13.95) | -3.23 (16.15) |
  Week 9: number analyzed (Participants) | 0 | 0 | 32
  Week 9 |  |  | -6.67 (17.19)
  Week 12: number analyzed (Participants) | 24 | 52 | 25
  Week 12 | -7.78 (13.57) | -5.10 (15.54) | -6.40 (16.61)
  Week 15: number analyzed (Participants) | 0 | 0 | 16
  Week 15 |  |  | -7.08 (14.90)
  Week 16: number analyzed (Participants) | 19 | 30 | 0
  Week 16 | -9.12 (17.10) | -5.11 (16.67) |
  Week 18: number analyzed (Participants) | 0 | 0 | 9
  Week 18 |  |  | -3.70 (14.95)
  Week 20: number analyzed (Participants) | 16 | 23 | 0
  Week 20 | -7.92 (19.51) | -0.87 (14.95) |
  Week 21: number analyzed (Participants) | 0 | 0 | 8
  Week 21 |  |  | -8.33 (17.37)
  Week 24: number analyzed (Participants) | 11 | 20 | 6
  Week 24 | -5.45 (9.81) | -3.00 (18.67) | 0.00 (16.87)
  Week 27: number analyzed (Participants) | 0 | 0 | 7
  Week 27 |  |  | 0.95 (15.60)
  Week 28: number analyzed (Participants) | 8 | 19 | 0
  Week 28 | -5.00 (9.92) | -3.16 (15.29) |
  Week 30: number analyzed (Participants) | 0 | 0 | 5
  Week 30 |  |  | -8.00 (20.76)
  Week 32: number analyzed (Participants) | 10 | 18 | 0
  Week 32 | -4.67 (11.35) | -10.74 (21.10) |
  Week 33: number analyzed (Participants) | 0 | 0 | 4
  Week 33 |  |  | -1.67 (13.74)
  Week 36: number analyzed (Participants) | 6 | 15 | 3
  Week 36 | -12.22 (14.25) | -1.78 (16.23) | 4.44 (15.40)
  Week 39: number analyzed (Participants) | 0 | 0 | 3
  Week 39 |  |  | 2.22 (19.25)
  Week 40: number analyzed (Participants) | 4 | 11 | 0
  Week 40 | -5.00 (11.39) | -0.61 (16.18) |
  Week 42: number analyzed (Participants) | 0 | 0 | 3
  Week 42 |  |  | 4.44 (15.40)
  Week 44: number analyzed (Participants) | 4 | 14 | 0
  Week 44 | 1.67 (3.33) | 3.33 (16.07) |
  Week 45: number analyzed (Participants) | 0 | 0 | 3
  Week 45 |  |  | 4.44 (15.40)
  Week 48: number analyzed (Participants) | 3 | 11 | 2
  Week 48 | -13.33 (6.67) | 1.82 (9.47) | 0.00 (18.86)
  Week 51: number analyzed (Participants) | 0 | 0 | 2
  Week 51 |  |  | 0.00 (18.86)
  Week 52: number analyzed (Participants) | 4 | 11 | 0
  Week 52 | -5.00 (6.38) | 3.64 (10.05) |
  Week 54: number analyzed (Participants) | 0 | 0 | 2
  Week 54 |  |  | 0.00 (18.86)
  Week 56: number analyzed (Participants) | 3 | 8 | 0
  Week 56 | -2.22 (3.85) | 5.00 (13.69) |
  Week 57: number analyzed (Participants) | 0 | 0 | 2
  Week 57 |  |  | 0.00 (18.86)
  Week 60: number analyzed (Participants) | 2 | 9 | 2
  Week 60 | -3.33 (4.71) | 2.96 (11.60) | 0.00 (18.86)
  Week 64: number analyzed (Participants) | 2 | 5 | 0
  Week 64 | -6.67 (18.86) | -2.67 (10.11) |
  Week 68: number analyzed (Participants) | 0 | 1 | 0
  Week 68 |  | 0.00 (0.00) |
  Treatment Discontinuation: number analyzed (Participants) | 40 | 66 | 39
  Treatment Discontinuation | -17.00 (19.21) | -16.24 (23.49) | -11.79 (19.01)
  Long Term Follow Up Month 3: number analyzed (Participants) | 9 | 15 | 11
  Long Term Follow Up Month 3 | -22.29 (24.29) | -15.11 (16.80) | -20.00 (26.67)
  Long Term Follow Up Month 6: number analyzed (Participants) | 9 | 10 | 5
  Long Term Follow Up Month 6 | -14.07 (17.14) | -10.00 (14.14) | -8.00 (15.92)
  Long Term Follow Up Month 30: number analyzed (Participants) | 0 | 1 | 1
  Long Term Follow Up Month 30 |  | -20.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available. | 13.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available.
  Long Term Follow Up Month 33: number analyzed (Participants) | 0 | 1 | 1
  Long Term Follow Up Month 33 |  | -20.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available. | 13.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available.
  Long Term Follow Up Month 36: number analyzed (Participants) | 0 | 1 | 1
  Long Term Follow Up Month 36 |  | -20.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available. | 13.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available.

6. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life-C30 Questionnaire (EORTC QLQ-C30) Global Quality of Life Sub-scale Score at the End of the Study
Description: as for outcome 5
Time Frame: Baseline, end of the study (up to approximately 2.5 years)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units of a scale
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
Number analyzed (Participants) | 57 | 125 | 61
units of a scale
  Week 3: number analyzed (Participants) | 0 | 0 | 49
  Week 3 |  |  | -1.70 (17.76)
  Week 4: number analyzed (Participants) | 44 | 100 | 0
  Week 4 | -6.44 (18.84) | -7.00 (21.24) |
  Week 6: number analyzed (Participants) | 0 | 0 | 48
  Week 6 |  |  | -4.86 (17.43)
  Week 8: number analyzed (Participants) | 29 | 78 | 0
  Week 8 | -8.05 (15.98) | -4.38 (22.58) |
  Week 9: number analyzed (Participants) | 0 | 0 | 31
  Week 9 |  |  | -4.84 (15.78)
  Week 12: number analyzed (Participants) | 24 | 51 | 25
  Week 12 | -1.04 (18.60) | -4.25 (18.51) | -3.67 (15.42)
  Week 15: number analyzed (Participants) | 0 | 0 | 16
  Week 15 |  |  | -4.69 (12.16)
  Week 16: number analyzed (Participants) | 20 | 30 | 0
  Week 16 | -4.39 (18.08) | -1.94 (23.64) |
  Week 18: number analyzed (Participants) | 0 | 0 | 9
  Week 18 |  |  | 7.41 (18.37)
  Week 20: number analyzed (Participants) | 16 | 23 | 0
  Week 20 | 0.52 (18.38) | 4.71 (23.28) |
  Week 21: number analyzed (Participants) | 0 | 0 | 8
  Week 21 |  |  | 6.25 (19.29)
  Week 24: number analyzed (Participants) | 11 | 20 | 6
  Week 24 | -3.79 (20.19) | 3.75 (23.95) | -6.94 (19.31)
  Week 27: number analyzed (Participants) | 0 | 0 | 7
  Week 27 |  |  | -2.38 (19.07)
  Week 28: number analyzed (Participants) | 8 | 19 | 0
  Week 28 | -8.33 (17.25) | 0.00 (31.18) |
  Week 30: number analyzed (Participants) | 0 | 0 | 5
  Week 30 |  |  | 5.00 (15.14)
  Week 32: number analyzed (Participants) | 10 | 18 | 0
  Week 32 | -5.00 (14.80) | 1.39 (23.79) |
  Week 33: number analyzed (Participants) | 0 | 0 | 4
  Week 33 |  |  | 6.25 (17.18)
  Week 36: number analyzed (Participants) | 6 | 15 | 3
  Week 36 | 0.00 (7.45) | 5.56 (16.86) | 16.67 (25.00)
  Week 39: number analyzed (Participants) | 0 | 0 | 3
  Week 39 |  |  | 22.22 (17.35)
  Week 40: number analyzed (Participants) | 4 | 11 | 0
  Week 40 | 2.08 (10.49) | 11.36 (12.51) |
  Week 42: number analyzed (Participants) | 0 | 0 | 3
  Week 42 |  |  | 25.00 (16.67)
  Week 44: number analyzed (Participants) | 4 | 14 | 0
  Week 44 | 0.00 (13.61) | 9.52 (15.63) |
  Week 45: number analyzed (Participants) | 0 | 0 | 3
  Week 45 |  |  | 19.44 (9.62)
  Week 48: number analyzed (Participants) | 3 | 11 | 2
  Week 48 | -2.78 (4.81) | 10.61 (15.85) | 8.33 (0.00)
  Week 51: number analyzed (Participants) | 0 | 0 | 2
  Week 51 |  |  | 8.33 (0.00)
  Week 52: number analyzed (Participants) | 4 | 11 | 0
  Week 52 | 4.17 (15.96) | 12.12 (17.62) |
  Week 54: number analyzed (Participants) | 0 | 0 | 2
  Week 54 |  |  | 12.50 (5.89)
  Week 56: number analyzed (Participants) | 3 | 8 | 0
  Week 56 | -5.56 (9.62) | 18.75 (9.71) |
  Week 57: number analyzed (Participants) | 0 | 0 | 2
  Week 57 |  |  | 8.33 (0.00)
  Week 60: number analyzed (Participants) | 2 | 9 | 2
  Week 60 | -4.17 (17.68) | 16.67 (15.59) | 8.33 (0.00)
  Week 64: number analyzed (Participants) | 2 | 5 | 0
  Week 64 | -4.17 (5.89) | 6.67 (24.58) |
  Week 68: number analyzed (Participants) | 0 | 1 | 0
  Week 68 |  | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available. |
  Treatment Discontinuation: number analyzed (Participants) | 39 | 66 | 39
  Treatment Discontinuation | -19.87 (23.93) | -14.27 (25.98) | -14.53 (20.48)
  Long Term Follow-up Month 3: number analyzed (Participants) | 9 | 15 | 11
  Long Term Follow-up Month 3 | -21.30 (28.60) | -6.11 (22.15) | -11.36 (20.16)
  Long Term Follow-up Month 6: number analyzed (Participants) | 9 | 10 | 5
  Long Term Follow-up Month 6 | -13.89 (19.09) | -15.83 (15.44) | -11.67 (15.14)
  Long Term Follow-up Month 30: number analyzed (Participants) | 0 | 1 | 1
  Long Term Follow-up Month 30 |  | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available. | 8.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available.
  Long Term Follow-up Month 33: number analyzed (Participants) | 0 | 1 | 1
  Long Term Follow-up Month 33 |  | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available. | 8.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available.
  Long Term Follow-up Month 36: number analyzed (Participants) | 0 | 1 | 1
  Long Term Follow-up Month 36 |  | 0.00 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available. | 8.33 (NA) — The standard deviation is a measure of the amount of variation or dispersion of a set of values. Number analyzed is 1 so SD is not available.

7. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Baseline, end of the study (up to approximately 2.5 years)
Population: Analysis was performed on the SAF population.
Measure: Number; unit: percentage of participants
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
Number analyzed (Participants) | 80 | 179 | 90
percentage of participants
  Serious AEs | 23.8 | 39.7 | 16.7
  Non-serious AEs | 97.5 | 97.8 | 93.3

8. Secondary Outcome: Plasma Concentration of Cobimetinib
Time Frame: Predose (0 hours) and 3 to 6 hours after dose on Day 15 of Cycles 1 and 4 (1 cycle = 28 days) (up to approximately 2.5 years).
Population: The pharmacokinetic (PK) evaluable population included all participants who received any dose of study medication and who had at least one post-baseline PK sample available. Only included participants in the Cobimetnib arm
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Cobimetinib + Atezolizumab
Number analyzed (Participants) | 124
Nanogram/milliliter (ng/mL)
  Cycle 1 Day 15 - Predose | 195 (190.0)
  Cycle 1 Day 15 - Postdose: number analyzed (Participants) | 122
  Cycle 1 Day 15 - Postdose | 362 (89.4)
  Cycle 4 Day 15 - Predose: number analyzed (Participants) | 51
  Cycle 4 Day 15 - Predose | 94.3 (741.9)
  Cycle 4 Day 15 - Postdose: number analyzed (Participants) | 44
  Cycle 4 Day 15 - Postdose | 210 (273.4)

9. Secondary Outcome: Serum Concentration of Atezolizumab
Description: Pre-infusion (0 hours) on Day 1 of Cycles 1 to 4; 30 minutes post-infusion on Day 1 of Cycles 1 and 4; pre-infusion (0 hours) on Day 1 of Cycle 8 and every 8 cycles thereafter; at treatment discontinuation; 120 days after treatment discontinuation (up to approximately 2.5 years) (1 cycle = 28 days)
Time Frame: Pre-infusion (0 hours) on Day 1 of Cycle 1 up to approximately 2.5 years. Detailed time frame is explained in the outcome measure description field.
Population: The pharmacokinetic (PK) evaluable population included all participants who received any dose of study medication and who had at least one post-baseline PK sample available. Also, only included participants to whom Atezolizumab was administered.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Arm/Group | Atezolizumab | Cobimetinib + Atezolizumab
Number analyzed (Participants) | 89 | 179
microgram/milliliter (ug/mL)
  Cycle 1 Day 1 - Predose: number analyzed (Participants) | 84 | 176
  Cycle 1 Day 1 - Predose | NA (NA) — If more than one-third values were less than reportable, then only the median and maximum are reported and other summary statistics are displayed as non-reportable. | NA (NA) — If more than one-third values were less than reportable, then only the median and maximum are reported and other summary statistics are displayed as non-reportable.
  Cycle 1 Day 1 - 30 min post dose: number analyzed (Participants) | 81 | 164
  Cycle 1 Day 1 - 30 min post dose | 348 (150.0) | 259 (141.0)
  Cycle 2 Day 1 - Predose: number analyzed (Participants) | 73 | 139
  Cycle 2 Day 1 - Predose | 81.5 (35.7) | 68.2 (191.2)
  Cycle 2 Day 1 - 30 min post dose: number analyzed (Participants) | 1 | 0
  Cycle 2 Day 1 - 30 min post dose | 56.2 (NA) — The amount of variation is not available as the number analyzed is 1. |
  Cycle 3 Day 1 - Predose: number analyzed (Participants) | 65 | 85
  Cycle 3 Day 1 - Predose | 118 (45.4) | 133 (51.2)
  Cycle 4 Day 1 - Predose: number analyzed (Participants) | 37 | 65
  Cycle 4 Day 1 - Predose | 146 (52.4) | 167 (48.4)
  Cycle 4 Day 1 - 30 min post dose: number analyzed (Participants) | 35 | 57
  Cycle 4 Day 1 - 30 min post dose | 487 (41.5) | 415 (37.2)
  Cycle 5 Day 1 - Predose: number analyzed (Participants) | 1 | 0
  Cycle 5 Day 1 - Predose | 155 (NA) — The amount of variation is not available as the number analyzed is 1. |
  Cycle 5 Day 1 - 30 min post dose: number analyzed (Participants) | 1 | 0
  Cycle 5 Day 1 - 30 min post dose | 456 (NA) — The amount of variation is not available as the number analyzed is 1. |
  Cycle 8 Day 1 - Predose: number analyzed (Participants) | 11 | 22
  Cycle 8 Day 1 - Predose | 138 (54.6) | 198 (52.6)
  Cycle 16 Day 1 - Predose: number analyzed (Participants) | 3 | 1
  Cycle 16 Day 1 - Predose | 226 (24.4) | 264 (NA) — The amount of variation is not available as the number analyzed is 1.
  Treatment Discontinuation: number analyzed (Participants) | 49 | 102
  Treatment Discontinuation | 97.9 (114.5) | 76.6 (184.9)
  Unscheduled: number analyzed (Participants) | 18 | 27
  Unscheduled | 0.784 (2159.5) | 0.539 (NA) — If more than one-third values were less than reportable, then only the median and maximum are reported and other summary statistics are displayed as non-reportable.

10. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Atezolizumab
Time Frame: Pre-infusion (0 hours) on Day 1 of Cycles 1 to 4, 8, and every 8 cycles thereafter; at treatment discontinuation; 120 days after treatment discontinuation (up to approximately 2.5 years) (1 cycle = 28 days)
Population: Analysis was performed on the SAF population and included participants with at least one predose and one postdose ATA assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Cobimetinib + Atezolizumab | Atezolizumab
Number analyzed (Participants) | 160 | 80
percentage of participants | 43.8 | 41.3

ADVERSE EVENTS:
Time Frame: From baseline to end of study (approximately 2.5 years).
Description: ITT was monitored for All-Cause Mortality, the safety analysis set (SAF) was assessed for Serious Adverse Events and Other (Not Including Serious) Adverse Events. SAF included all enrolled participants who received at least one dose of any study medication.
Arm/Group | Regorafenib | Cobimetinib + Atezolizumab | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 62/90 | 136/183 | 72/90
Serious Adverse Events (participants affected / at risk) | 19/90 | 71/183 | 15/90
Other Adverse Events (participants affected / at risk) | 78/80 | 173/179 | 81/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Regorafenib (N=90) | Cobimetinib + Atezolizumab (N=183) | Atezolizumab (N=90)
ANAEMIA (Blood and lymphatic system disorders) | 0/80 (0) | 5/179 (5) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
MACULOPATHY (Eye disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2/80 (2) | 2/179 (2) | 1 (1)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0/80 (0) | 2/179 (2) | 1 (1)
COLONIC FISTULA (Gastrointestinal disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3/80 (3) | 6/179 (6) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1/80 (1) | 1/179 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 2/80 (2) | 1/179 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0/80 (0) | 0/179 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0/80 (0) | 0/179 (0) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
VOLVULUS OF SMALL BOWEL (Gastrointestinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1/80 (1) | 1/179 (1) | 0 (0)
ASTHENIA (General disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
CHILLS (General disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
DEATH (General disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
FATIGUE (General disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
INFLAMMATION (General disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
PYREXIA (General disorders) | 3/80 (3) | 12/179 (15) | 2 (2)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0/80 (0) | 0/179 (0) | 1 (1)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0/80 (0) | 0/179 (0) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 0/80 (0) | 1/179 (2) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 0/80 (0) | 0/179 (0) | 1 (1)
ABDOMINAL HERNIA INFECTION (Infections and infestations) | 0/80 (0) | 0/179 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
BACTERIAL SEPSIS (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
INFECTION (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
LUNG INFECTION (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0/80 (0) | 2/179 (3) | 0 (0)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
PULMONARY SEPSIS (Infections and infestations) | 0/80 (0) | 1/179 (1) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1/80 (1) | 1/179 (1) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 0/80 (0) | 1/179 (1) | 0 (0)
SEPSIS (Infections and infestations) | 2/80 (2) | 4/179 (4) | 0 (0)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1/80 (1) | 0/179 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0/80 (0) | 2/179 (2) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0/80 (0) | 1/179 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0/80 (0) | 3/179 (3) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0/80 (0) | 1/179 (1) | 0 (0)
STOMA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0/80 (0) | 0/179 (0) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0/80 (0) | 2/179 (2) | 0 (0)
INFLUENZA A VIRUS TEST POSITIVE (Investigations) | 0/80 (0) | 1/179 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0/80 (0) | 1/179 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0/80 (0) | 0/179 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1/80 (1) | 2/179 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0/80 (0) | 0/179 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0/80 (0) | 2/179 (2) | 1 (1)
ATAXIA (Nervous system disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0/80 (0) | 2/179 (2) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
NONINFECTIVE ENCEPHALITIS (Nervous system disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0/80 (0) | 2/179 (2) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 0/80 (0) | 1/179 (1) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
NEPHRITIS (Renal and urinary disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
STERILE PYURIA (Renal and urinary disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1/80 (1) | 0/179 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0/80 (0) | 1/179 (2) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0/80 (0) | 1/179 (1) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0/80 (0) | 1/179 (1) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0/80 (0) | 1/179 (1) | 0 (0)
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 0/80 (0) | 0/179 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (N=80) | Cobimetinib + Atezolizumab (N=179) | Atezolizumab (N=90)
ANAEMIA (Blood and lymphatic system disorders) | 8 (9) | 25 (28) | 5 (5)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 10 (10) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 21 (27) | 30 (34) | 13 (19)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 3 (3) | 7 (8)
CONSTIPATION (Gastrointestinal disorders) | 17 (19) | 33 (41) | 11 (12)
DIARRHOEA (Gastrointestinal disorders) | 30 (59) | 115 (200) | 17 (23)
DRY MOUTH (Gastrointestinal disorders) | 4 (4) | 9 (9) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 10 (10) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 12 (13) | 67 (93) | 19 (23)
PROCTALGIA (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 13 (21) | 18 (18) | 0 (0)
VOMITING (Gastrointestinal disorders) | 9 (10) | 52 (79) | 13 (15)
ASTHENIA (General disorders) | 17 (22) | 37 (54) | 12 (19)
CHEST PAIN (General disorders) | 4 (4) | 5 (5) | 2 (2)
CHILLS (General disorders) | 4 (4) | 14 (15) | 4 (5)
FACE OEDEMA (General disorders) | 0 (0) | 10 (12) | 0 (0)
FATIGUE (General disorders) | 38 (46) | 65 (75) | 24 (28)
MUCOSAL INFLAMMATION (General disorders) | 6 (8) | 16 (19) | 4 (6)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 27 (32) | 8 (9)
PYREXIA (General disorders) | 20 (25) | 53 (67) | 12 (13)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (4) | 4 (6) | 6 (6)
URINARY TRACT INFECTION (Infections and infestations) | 4 (8) | 8 (10) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (6) | 10 (17) | 5 (5)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (8) | 16 (27) | 6 (8)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 14 (14) | 8 (11)
BLOOD BILIRUBIN INCREASED (Investigations) | 4 (7) | 3 (3) | 2 (2)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 3 (5) | 22 (39) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 5 (6) | 3 (3) | 0 (0)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 4 (4) | 3 (5) | 3 (3)
LIPASE INCREASED (Investigations) | 6 (7) | 9 (10) | 1 (2)
WEIGHT DECREASED (Investigations) | 17 (18) | 8 (9) | 7 (7)
DECREASED APPETITE (Metabolism and nutrition disorders) | 34 (40) | 49 (57) | 21 (27)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 5 (5) | 7 (7) | 2 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (4) | 14 (17) | 1 (1)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 7 (7) | 11 (11) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 14 (14) | 8 (8)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (10) | 17 (21) | 13 (15)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 2 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (10) | 9 (12) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (8) | 12 (16) | 6 (6)
DIZZINESS (Nervous system disorders) | 3 (3) | 10 (12) | 0 (0)
HEADACHE (Nervous system disorders) | 10 (12) | 17 (21) | 11 (11)
INSOMNIA (Psychiatric disorders) | 3 (3) | 9 (9) | 6 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 33 (35) | 12 (12)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 19 (27) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 36 (41) | 12 (12)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (8) | 2 (2)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2) | 46 (56) | 2 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 14 (14) | 3 (3)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3) | 0 (0)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 42 (70) | 3 (3) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 22 (25) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 17 (19) | 85 (122) | 8 (8)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 (3) | 11 (12) | 1 (1)
HYPERTENSION (Vascular disorders) | 25 (31) | 9 (10) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT02788279/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT02788279/SAP_001.pdf